CLINICAL TRIAL: NCT06707740
Title: Comparison of the Effect of Capsular Bend on the Rotational Stability Between Two Toric Intraocular Lenses
Status: Active, not recruiting | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: SSOCT-toric
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 AcrySof IQ(SN6AT) implantation after cataract surgery.
- Group 2TECNIS（ZCU） implantation after cataract surgery.

SUMMARY:
(1) To compare the difference of rotational stability and CBI between AcrySof IQ(SN6AT) and TECNIS(ZCU) after cataract surgery. (2) To evaluate the influence of capsular bending on the rotational stability of these two kinds of intraocular lenses.

DETAILED DESCRIPTION:
To compare the difference of rotational stability and CBI between AcrySof IQ(SN6AT) and TECNIS (ZCU) torus intraocular lenses implanted after cataract surgery, and analyze the influence of capsular bag bending on the rotational stability of two kinds of astigmatism correction intraocular lenses after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:1.The patient's age is over 18 years old. 2.Diagnosed as age-related cataract Corneal astigmatism measured before operation is > 0.75 D or predicted after operation after taking into account surgical astigmatism (SIA).

3.Pupil diameter > 7 mm after mydriasis. 4.The astigmatism meridian between IOLMaster and Pentacam is the same (the meridian difference between the two instruments is within 15).

5.After operation, the anterior capsule completely covered the edge of intraocular lens optical surface.

6.Able to understand, cooperate and complete all follow-up.

-

Exclusion Criteria:

1. Moderate and severe dry eye
2. There is irregular corneal astigmatism.
3. Combined with other ophthalmic diseases Previous history of ophthalmic surgery.
4. The capsulorhexis is too large or eccentric, which can not cover the optical zone of intraocular lens all around, and there are intraoperative or postoperative complications.

   -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Included in Eye Hospital of Wenzhou Medical University for "phacoemulsification combined with intraocular lens implantation"
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Capsular bend index | 1-2 hours after operation, 1 day, 1 week, 1 month and 3 months.
  The average value of the capsular bag bending stage in different positions of IOL represents the speed of the whole capsular bag bending formation in the eye.
IOL rotation degree | 1-2 hours after operation, 1 day, 1 week, 1 month and 3 months.
  The difference of degrees between the actually measured Toric IOL astigmatism axes at two adjacent follow-up time points.
Toric IOL total axial deviation | 1-2 hours after operation, 1 day, 1 week, 1 month and 3 months.
  The degree difference between the actual axial position and the target axial position of Toric IOL is different.

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology and Optometry Hospital, Wenzhou, Wenzhou, China

IPD SHARING:
Plan to Share IPD: No